CLINICAL TRIAL: NCT01810679
Title: Clinical Investigation of the Perceval S Sutureless Heart Valve
Brief Title: Perceval S Aortic Heart Valve Study- North America
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA approval
Sponsor: Sorin Group USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G120053
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Stenosis With Insufficiency; Regurgitation, Aortic Valve; Aortic Valve Incompetence
Keywords: aortic valve replacement; aortic stenosis; aortic steno-insufficiency; Perceval; Sutureless aortic heart valve
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Perceval S Aortic Heart Valve (Experimental): Treatment with the Perceval S Aortic Heart Valve
  Interventions: Device: Perceval S Aortic Heart Valve

INTERVENTIONS:
Device: Perceval S Aortic Heart Valve — Perceval S Sutureless Aortic Heart Valve

SUMMARY:
To demonstrate the safety and effectiveness of the Perceval S heart valve when used to replace a diseased or dysfunctional aortic valve or aortic valve prosthesis.

DETAILED DESCRIPTION:
This investigation is a prospective, non-randomized, multi-center trial of the PERCEVAL valve implanted in patients requiring aortic valve replacement. The study will be conducted in a maximum of 25 centers in the United States. Patients will be evaluated at each of the following time intervals:preoperative, at implant, in the early postoperative period, in the late postoperative period (between 3 and 6 months postoperatively), at 1 year (between 11 and 13 months postoperatively), and annually until study completion. The duration of the study is anticipated to be 5 years.

ELIGIBILITY:
Inclusion criteria:

1. Subjects of age >= 18 years.
2. Subjects with aortic valve stenosis or steno-insufficiency.
3. The subject is willing to sign the informed consent.
4. The subject in which preoperative evaluation indicated the need for native or prosthetic aortic valve replacement.
5. The subject is located in a geographic location that will enable the subject to return to the study site for all follow-up examinations (i.e. geographically stable).
6. Subject will be available to the investigator(s) for postoperative follow-up beyond one year.

Exclusion criteria:

1. The subject has preexisting valve prosthesis or annuloplasty ring in the mitral, pulmonic or tricuspid position.
2. The subject requires a double or multiple valve replacement or repair of the mitral, tricuspid, or pulmonic valve.
3. The subject has a previously implanted PERCEVAL valve that requires replacement.
4. Subjects requiring simultaneous cardiac procedures, apart from septal myectomy and/or coronary by-pass.
5. The subject has active endocarditis.
6. Subjects with active myocarditis
7. The subject is or will be participating in a concomitant research study of an investigational product.
8. Subjects with aneurysmal dilation or dissection of the ascending aortic wall.
9. The subject is a minor, drug abuser, alcohol abuser, prison inmate, institutionalized, or is unable to give informed consent.
10. The subject has a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy of less than 1 year, or the implant of the device produces an unacceptable increased risk to the patient.
11. Subjects with known hypersensitivity to nickel alloys.
12. The subject is undergoing renal dialysis for chronic renal failure or has hyperparathyroidism.
13. The subject has had an acute preoperative neurological deficit, myocardial infarction, or cardiac event that has not returned to baseline or stabilized ≥30 days prior to the planned valve implant surgery.
14. Subject is known to be noncompliant or is unlikely to complete the study.
15. Subjects with an aortic root enlargement, where the ratio between the diameter of the sino-tubular junction and the annulus diameter, assessed by TTE, is > 1.3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | One-year
  To demonstrate that the complication and survival rates for the PERCEVAL S valve are comparable to appropriate historical controls manifested as objective performance criteria (OPCs) and to that reported for other stented bioprostheses in the literature
Primary Efficacy Endpoint | One-year
  To demonstrate that the rate of valve success for the PERCEVAL S valve is comparable to that of appropriate historical controls

SECONDARY OUTCOMES:
Secondary Efficacy Outcomes | One-year
  To demonstrate that the hemodynamic performance of the PERCEVAL S valve is comparable to that reported in the literature for other stented aortic bioprostheses
Secondary Efficacy Outcomes | One-year
  To demonstrate clinically significant improvements in overall patient condition by comparison of preoperative and postoperative NYHA functional classifications
Secondary Efficacy Outcomes | One-year
  To demonstrate that the rate of device technical success for the PERCEVAL S valve is comparable to that of appropriate historical controls

OTHER OUTCOMES:
Supplementary Analyses | Discharge
  Rates of cross-clamp time, cardiopulmonary bypass time, length of stay in ICU, length of hospital, and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Suri, MD, DPhil, Principal Investigator — The Cleveland Clinic
Locations (21):
- United States (21):
  - East Alabama Medical Center, Opelika, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Colorado Denver, Aurora, Colorado
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Oakwood Hospital, Dearborn, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian - Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center/Albert Einstein College of Medicine, New York, New York
  - Lenox Hill/NS-LIJ, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cardiothoracic and Vascluar Surgeons, Austin, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - University of Washington, Seattle, Washington